CLINICAL TRIAL: NCT04518033
Title: Measuring Droplets in Children
Acronym: MeDiC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Peter Moschovis, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020P002630
Record Dates: First submitted 2020-08-12; First posted 2020-08-19 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Droplet Spread

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Face covering use (Experimental): Participants will be provided various commercially available face coverings
  Interventions: Device: Various commercially available face coverings

INTERVENTIONS:
Device: Various commercially available face coverings — Various commercially available face coverings

SUMMARY:
This study will measure the size and quantity of respiratory particle production in children under a variety of conditions, including face coverings/masks and various common activities.

ELIGIBILITY:
Inclusion Criteria:

- Age 3 to 17 years

Exclusion Criteria:

* Chronic neuromuscular conditions that affect respiration
* Tracheostomy tube
* Unable to wear a face mask

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2021-04-03 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
Respiratory particle production | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Peter P Moschovis, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No